CLINICAL TRIAL: NCT00489450
Title: Clinical Trial to Investigate the Influence of Alcohol on the Pharmacokinetics and Safety of SK3530 in Healthy Male Volunteers
Brief Title: Phase I Study to Investigate the Alcohol Interaction of SK3530
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SK3530_AI_2006
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-03

CONDITIONS: Erectile Dysfunction
Keywords: SK3530; alcohol; pharmacokinetics; safety
MeSH Terms: conditions — Erectile Dysfunction | interventions — 2-(5-(4-(2-hydroxyethyl)piperazin-1-ylsulfonyl)-2-n-propoxyphenyl)-5-ethyl-7-n-propyl-3,5-dihydro-4H-pyrrolo(3,2-d)pyrimidin-4-one dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SK3530

SUMMARY:
This study was designed to investigate the alcohol effect of SK3530 on the pharmacokinetics (PKs) and safety.

DETAILED DESCRIPTION:
This study was a randomized, open, single-dose, three-treatment, three-period, three-sequence, crossover study in which subjects were received, in random order, SK3530 100mg alone, 0.5g/Kg of alcohol alone, and SK3530 plus alcohol together. There was a minimum of a 7 day washout period between treatments. The alcohol was diluted to 240 mL with water. The contents were drunk in 1 minutes or less. For SK3530 and metabolite measurement, plasma samples were collected at pre-scheduled time and the safety was monitored all through the study.

ELIGIBILITY:
Inclusion Criteria:

* ages 20 to 50
* body weight of IBM ± 20%

Exclusion Criteria:

* cardiovascular disease
* color-blindness or weakness
* no availability to intake 0.5 g/Kg alcohol
* abnormal supine blood preesure

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
PK parameters - AUC, Cmax | 24hr after administration

SECONDARY OUTCOMES:
Safety (Vital signs, Adverse events) | until post-study visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea